CLINICAL TRIAL: NCT00857636
Title: Better Breast and Cervical Cancer Control for Korean American Women
Brief Title: Behavioral Intervention Study for Better Breast and Cervical Cancer Control for Korean American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hae-Ra Han, Associate professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01CA129060 (NIH)
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer; Cervical Cancer
Keywords: Ethnic minority women; Cancer screening; Health literacy; Behavioral intervention; Breast Cancer screening; Cervical Cancer screening
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms | interventions — Health Literacy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Health Literacy (Experimental)
  Interventions: Behavioral: Health literacy, health message

INTERVENTIONS:
Behavioral: Health literacy, health message — The intervention will consist of three main components: (1) 2-hour in-class health literacy-focused education; (2) tailored telephone counseling; and (3) healthcare system navigation assistance tailored to the woman's specific barriers.

SUMMARY:
The long-term goal of this study is to build a sustainable,community-based outreach program using Korean American community health workers (CHWs) to promote breast and cervical screening among Korean American women, thereby reducing related morbidity and mortality. The study is designed to determine the effectiveness of a health literacy-focused tailored breast and cervical cancer control intervention delivered by CHWs.

The investigators hypothesized that, compared to KA women in the delayed intervention group, KA women who receive a health literacy-focused CHW intervention will demonstrate: (1) higher levels of adherence to screening for breast and cervical cancer, (2) greater levels of health literacy, (3) higher levels of breast and cervical cancer knowledge, and (4) improve decisional balance.

DETAILED DESCRIPTION:
Despite considerable progress in U.S. cancer control over the past 20 years, certain ethnic minority groups continue to experience significant health disparities. Recent immigrants including Korean Americans (KA), face an unequal cancer burden related to the significant language and cultural barriers they face in attempting to navigate the U.S. healthcare system. KA women have the second highest incidence of cervical cancer nationally and are experiencing rapid increases in breast cancer incidence. Not only are their breast and cervical cancers diagnosed at significantly later stages than those of whites, but they are also the least likely racial/ethnic group to receive early breast and cervical cancer screening.

This community-based behavioral intervention is designed 1) to evaluate, in a randomized controlled trial, the effects of our health literacy-focused cancer control intervention, delivered by trained CHWs, on the primary outcomes: mammography and Papanicolaou(Pap)test screening adherence, in a sample of 360 KA women, 2)to test the effects of the proposed intervention on the secondary outcomes: level of health literacy, breast and cervical knowledge, and decisional balance, in the KA sample.

ELIGIBILITY:
Inclusion Criteria:

1. age 21-65 years
2. self-identified as a KA woman
3. no mammogram and Pap test within the last 18 months
4. able to read and write Korean or English
5. willing to provide written study consent
6. willingness to provide written consent to allow the researchers to audit medical records for mammography and Pap test use.

Exclusion Criteria:

1. Potential participants with a cancer diagnosis, an acute and/or terminal condition
2. Psychiatric diagnosis (e.g., schizophrenia or cognitive impairment), or other conditions
3. Women who have undergone hysterectomy

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of participants who adhere to mammography and Papanicolaou(Pap) test screening guidelines | 6 months
  The primary outcome variables are self-reported receipt of, or intention to obtain mammography and/or Pap test. Self-reported intention as an outcome variable has been a common practice in the screening literature, since it has been found to be the best predictor of actual screening behavior.Number of participants who adhere to mammography and Pap test during 6 months period will be the primary outcomes.

SECONDARY OUTCOMES:
Health belief score about breast & cervical cancer | 6 months
  Secondary outcome variables include satisfaction with community health worker-led education sessions and follow-up, changes in other screening behaviors including clinical breast exam and breast self-exam, and breast, cervical cancer relevant health beliefs and knowledge. Health belief score will be assessed at baseline, 3, 6 months.
Knowledge score about breast & cervical cancer | 6 months
  Secondary outcome variables include satisfaction with community health worker-led education sessions and follow-up, changes in other screening behaviors including clinical breast exam and breast self-exam, and breast, cervical cancer relevant health beliefs and knowledge.Health knowledge score will be assessed at baseline, 3, 6 months.
Satisfaction score with community health worker-led intervention activities | 6 month follow-up
  Community health worker-led intervention activities include heatlh literacy focused structured education, monthly telephone counselings and other navigation activities to encourage the study participants to have mammogram and pap test. Satisfaction score will be measured at 6 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Hae-Ra Han, PhD, Principal Investigator — Johns Hopkins University, School of Nursing
Locations (1):
- Korean Resource Center, Ellicott City, Maryland, United States

REFERENCES:
- [Derived] Kim K, Kim S, Gallo JJ, Nolan MT, Han HR. Decision making about Pap test use among Korean immigrant women: A qualitative study. Health Expect. 2017 Aug;20(4):685-695. doi: 10.1111/hex.12507. Epub 2016 Sep 30. PMID 27687295
- [Derived] Choi E, Heo GJ, Song Y, Han HR. Community Health Worker Perspectives on Recruitment and Retention of Recent Immigrant Women in a Randomized Clinical Trial. Fam Community Health. 2016 Jan-Mar;39(1):53-61. doi: 10.1097/FCH.0000000000000089. PMID 26605955
- [Derived] Kim J, Huh BY, Han HR. Correlates of misperception of breast cancer risk among Korean-American Women. Women Health. 2016 Aug-Sep;56(6):634-49. doi: 10.1080/03630242.2015.1118722. Epub 2015 Nov 18. PMID 26580449
- [Derived] Schuster AL, Frick KD, Huh BY, Kim KB, Kim M, Han HR. Economic evaluation of a community health worker-led health literacy intervention to promote cancer screening among Korean American women. J Health Care Poor Underserved. 2015 May;26(2):431-40. doi: 10.1353/hpu.2015.0050. PMID 25913341
- [Derived] Han HR, Huh B, Kim MT, Kim J, Nguyen T. Development and validation of the assessment of health literacy in breast and cervical cancer screening. J Health Commun. 2014;19 Suppl 2(0 2):267-84. doi: 10.1080/10810730.2014.936569. PMID 25315598